CLINICAL TRIAL: NCT02133469
Title: Effectiveness of PCV7 in the Prevention of Nasopharyngeal Carriage of Vaccine Serotype (VT) Streptococcus Pneumoniae in 2 to 5 Years Old Healthy Chinese Children.
Brief Title: PCV7 in the Prevention of Nasopharyngeal Carriage of Vaccine Serotype (VT) Streptococcus Pneumoniae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Beijing Municipal Health Bureau (Other); Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Principal Investigator, Wu Jiang, Department of Immunization & Prevention,Beijing Center for Disease Control and Prevention, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BJCDCWJ201201
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Streptococcal Pneumonia; Nasopharyngeal Diseases; Vaccination Adverse Event
Keywords: Effectiveness; Prevenar; nasopharyngeal carriage; vaccine serotype
MeSH Terms: conditions — Pneumonia; Nasopharyngeal Diseases | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine; HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCV7 (Vaccine) (Experimental): Randomized group of 1634 subjects to be administered a single dose of PCV7 (Hib vaccine offered at end of study).
  Interventions: Biological: PCV7 (Pneumococcal 7-Valent Conjugate Vaccine)
- Hib vaccine (Active Comparator): Randomized group of 1634 subjects to be administered a single dose of Hib Vaccine(PCV7 vaccine offered at end of study).
  Interventions: Biological: Hib Vaccine

INTERVENTIONS:
Biological: PCV7 (Pneumococcal 7-Valent Conjugate Vaccine) — injection 0.5 mL, single dose
  Other Names: Prevenar
  Arms: PCV7 (Vaccine)
Biological: Hib Vaccine — Single Dose
  Arms: Hib vaccine

SUMMARY:
A parallel-group, randomized, open-label study will be performed in subjects receiving PCV7 and subjects receiving controlled vaccine Hib vaccine, to claim the efficacy of PCV7 in the prevention of NP carriage of vaccine-serotype S. pneumoniae (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F combined) in 2 to 5 years old healthy Chinese children.

DETAILED DESCRIPTION:
In 2005, clinical trials with PCV7 (Prevenar) were first conducted in China. In the phase 3 study involving Chinese infants, Prevenar was shown to be immunogenic, well tolerated, and safe when given either separately or concomitantly with a diphtheria, tetanus, and acellular pertussis (DTaP) vaccine at 3, 4, and 5 months of age. Controlled clinical trials elsewhere in the world showed the correlation between immunogenicity and disease prevention. In addition to the direct effect of Prevenar, immunization of children has also reduced the incidence of disease in adults. The changes are presumed to be due to reductions in nasopharyngeal carriage of vaccine serotype S. pneumoniae in children who have been vaccinated.

The purpose of this study will be to assess the effectiveness of Prevenar vaccination to reduce vaccine serotype (VT) NPC rates in Chinese children aged 2 to 5 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy children aged 2 to 5 years.
2. Evidence of a personally signed and dated informed consent document indicating that the parent(s) (or legal guardian) has been informed of all pertinent aspects of the study.
3. Subjects and parents / legal guardian/ adult caregiver who are willing and able to comply with scheduled visits, treatment plan, and other study procedures.
4. Available for entire study period and whose parent/legal guardian/adult caregiver can be reached by telephone.
5. Healthy child as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. Receipt of a full series or catch-up dose of licensed or investigational Hib vaccinations.
3. Contraindication to vaccination with a pneumococcal conjugate vaccine or Hib.
4. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
5. Known or suspected immune deficiency or suppression including treatment with systemic steroids, anti-metabolites, chemotherapy and immunomodulatory agents.
6. Major known congenital malformation or serious chronic disorder.
7. Malformation or injury of the nasopharynx that makes the procedure of taking a nasopharyngeal swab impossible.
8. Significant neurologic disorder including congenital neurological disease in sibling of the subject or history of seizure including febrile seizure, or significant stable or evolving disorder such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorder. Does not include resolving syndromes due to birth trauma such as Erb's palsy.
9. Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies) within 12 weeks prior to enrollment.
10. Participation in another investigational or interventional trial within the 28-day period before enrollment and during the conduct of the study. Participation in purely observational studies is acceptable.
11. Subjects whose parents or legal representative are investigational site staff members or subjects whose parents or legal representative are Pfizer employees directly involved in the conduct of the trial.

Temporary Exclusion Criteria(The following conditions are temporary or self-limiting and a subject may be included in the study once the condition(s) has/have resolved and no other exclusion criteria are met):

1. Subjects with current febrile illness (axillary temperature of ≥ 38.0ºC).
2. Subjects who used antibiotics within the previous 15 days.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3281 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Carriage Rate of Vaccine-Serotype S. pneumoniae at 180days after vaccination | 6 months

SECONDARY OUTCOMES:
Carriage Rate of vaccine-serotype S. pneumoniae in PCV7 group versus Hib group. | 60 days
Carriage rate of non-vaccine serotype S. pneumoniae in PCV7 group versus Hib group. | Baseline before vaccination
Carriage rate of non-vaccine serotype S. pneumoniae in PCV7 group versus Hib group. | 60 days after vaccination
Carriage rate of non-vaccine serotype S. pneumoniae in PCV7 group versus Hib group. | 6 months after vaccination
Carriage rate of individual serotype S. pneumoniae in PCV7 group and Hib group. | Baseline before vaccination
Carriage rate of individual serotype S. pneumoniae in PCV7 group and Hib group. | 60 days after vaccination
Carriage rates of individual serotype S. pneumoniae in PCV7 group and Hib group. | 6 months after vaccination
Carriage rate of antibiotic resistant S. pneumoniae as a group in PCV7 group and Hib group. | 6 months after vaccination
Percentage of adverse event related to vaccination in PVC7 group and Hib group. | 6 months after vaccination
Category of adverse event related to vaccination in PVC7 group and Hib group. | 6 months after vaccination
  Adverse effects are classified as referenced from the China Food and Drug Administration's "Preventive Vaccines Clinical Study Adverse Effects Assessment Standards". This evaluation of systemic reactions is partially based on standards for classification set by the United States National Institutes of Health and the National Institute of Allergy and Infectious Diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Jiang, Bachelor, Principal Investigator — Beijing Centers for Disease Control and Prevention
Locations (9):
- China (9):
  - Huairou District Center for Disease Prevention and Control, Beijing, Beijing Municipality
  - Daxing District Center for Disease Prevention and Control, Beijing, Beijing Municipality
  - Chongwen District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Shijingshan District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Xuanwu District Center for Disease Control and Prevention, Beijing, Beijing Municipality
  - Chaoyang District Center for Disease Control and Prevention, Chaoyang District, Beijing Municipality
  - Dongcheng District Center for Disease Control and Prevention, Dongcheng District, Beijing Municipality
  - Fengtai District Center for Disease Control and Prevention, Fengtai District, Beijing Municipality
  - Xicheng District Center for Disease Prevention and Control, Xicheng District, Beijing Municipality